CLINICAL TRIAL: NCT05783895
Title: Comparison of Pre-test Probability Model for Heparin-induced Thrombocytopenia in Post-operative Cardiac Surgery With Bypass Surgery
Brief Title: Comparison of Pre-test Probability Model for Heparin-induced Thrombocytopenia in Post-operative Cardiac Surgery
Acronym: TicTac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI190
Record Dates: First submitted 2023-03-09; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Heparin-induced Thrombocytopenia
Keywords: Cardiopulmonary Bypass; pre-test probability model

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed HIT: Comprehensive collection of patients with suspected and then proven HIT postoperatively from cardiac surgery with bypass surgery during the inclusion period.
  Interventions: Diagnostic Test: Post screening diagnostic test
- Absence of HIT: Patients with suspected and unconfirmed HIT postoperatively from cardiac surgery under CEC during the inclusion period.
  Interventions: Diagnostic Test: Post screening diagnostic test

INTERVENTIONS:
Diagnostic Test: Post screening diagnostic test — 1) anti-PF4/heparin antibody test (ELISA) and 2) in vitro platelet aggregation tests. The diagnosis of HIT is made when both tests are positive or when a platelet aggregation test is positive.

SUMMARY:
Heparin-induced thrombocytopenia (HIT) is a pro-thrombotic immunological condition that occurs in some patients exposed to heparin. The incidence of HIT is estimated at 0.1 to 0.3% of patients exposed to heparin, and rises to 3% in postoperative cardiac surgery. Cardiac surgery under CEC requires the use of high doses of heparin, which contributes to the increased incidence of HIT in this population. This high incidence is also explained by the comorbid profile of cardiac surgery patients, who often present risk factors for HIT (perioperative context, atrial fibrillation, organ failure, previous exposure to heparin, etc.). When it occurs postoperatively in cardiac surgery, there is a 28% increase in mortality, a 50% increase in morbidity, and an increase in hospitalization costs and length of stay. Although usually detected in medical wards on the basis of probability scores (4T, HEP), its diagnosis is less easy in postoperative cardiac surgery. Because of the many differential diagnoses, the screening scores usually used are less effective, and HIT is often diagnosed late, in patients who may have already developed a thromboembolic complication, which sometimes proves fatal. In addition, the diagnostic tests for HIT are compromised and lose their sensitivity in postoperative cardiac surgery, given the high incidence of seroconversion observed after extracorporeal circulation. Indeed, more than 50% of patients have antibodies to PF4/heparin, but only 1 to 2% of them have true HIT.These elements highlight the need to develop effective screening scores for HIT in postoperative cardiac surgery, given the complications to which patients are exposed in the event of underdiagnosis but also in the event of overdiagnosis. Other screening scores are being studied, not yet validated in cardiac surgery, such as the CPB score or the GFHT score. Early recognition of HIT would reduce the morbidity and mortality associated with this condition.

The present study should make it possible to identify the most effective HIT probability score among those used in routine screening and thus to orient towards screening for this condition as early as possible, and consequently reduce the associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Major patients, who underwent cardiac surgery with cardiopulmonarybypass between 01/01/2010 and 12/31/2021, in whom HIT was suspected postoperatively.

Exclusion Criteria:

* Patients with known preoperative HIT,
* cardiac surgery patients without bypass surgery,
* diagnostic tests for HIT not performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study concerns patients over 18 years of age, undergoing scheduled or emergency cardiac surgery with postoperative thrombocytopenia and suspected HIT.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the intrinsic performance of HIT tests | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To compare the intrinsic performance (sensitivity, specificity) of 4 HIT screening scores (4T, HET, GFHT, CPB) in postoperative cardiac surgery under CEC.

SECONDARY OUTCOMES:
Evaluation of the extrinsic performance of HIT tests | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To compare the extrinsic performance (sensitivity, specificity) of 4 HIT screening scores (4T, HET, GFHT, CPB) in postoperative cardiac surgery under CEC.
30-day postoperative mortality | between the date of confirmation of HIT and 30 days from the date of hospitalization
  To estimate 30-day postoperative mortality of cardiac surgery under CEC in patients with confirmed HIT.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas KLEIN, MD, Study Director — Nancy Hospital
Locations (1):
- 'CHRU Nancy, Vandœuvre-lès-Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: No